CLINICAL TRIAL: NCT00453531
Title: Pilot Study for the Development of Transient Forearm Endothelial Dysfunction
Brief Title: Model System for Transient Forearm Blood Vessel Dysfunction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Michael Sack, M.D./National Heart, Lung and Blood Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 070124; 07-H-0124
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2022-08-09 (Actual); Status verified 2009-02

CONDITIONS: Limb Ischemia; Ischemic Preconditioning
Keywords: Forearm Ischemia; Endothelial Function; Acetyicholine Vasodilation; Venous Plethysmography; Healthy Volunteer; HV
MeSH Terms: interventions — Acetylcholine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteers (Experimental)
  Interventions: Procedure: Limb Ischemia; Drug: Acetylcholine

INTERVENTIONS:
Procedure: Limb Ischemia
Drug: Acetylcholine

SUMMARY:
This study will develop a model system that can be used to test medications for improving the ability of blood vessels to resist damage from diseases such as heart attack and stroke. The endothelium (inner layer of blood vessels) has built-in defense mechanisms to prevent blockage of blood flow, including the ability to stretch the vessel when it senses that blood flow is threatened. People with heart attack risk factors, such as high cholesterol, smoking and diabetes lose this ability. This study will develop a model that can measure the response to a lack of blood flow in the arm and be used to test new medicines to improve blood vessel health.

Healthy males between 18 and 45 years of age who have no history of high blood pressure, high cholesterol, or diabetes and who have not smoked for at least 3 months before entering the study may be eligible to enroll.

Participants lie in an adjustable reclining bed. Small catheters (tubes) are placed in the artery and vein of the forearm of the non-dominant arm at the inside of the elbow. Blood samples are collected from the tubes. Then, pressure cuffs are placed on both wrists and upper arms. A strain gauge (rubber band-type device) is placed around the forearms. The pressure cuffs are inflated and blood flows into the forearm, stretching the strain gauge at a rate proportional to the blood flow. Then, small doses of acetylcholine (a medicine that causes blood vessels to expand) are injected into the artery tube. After 20 minutes, blood flow to the non-dominant arm is blocked by inflating the pressure cuff. The subject squeezes a rubber ball about every 2 seconds for 90 seconds. The cuff is deflated after 15 minutes and blood samples are withdrawn from the tube in the vein. After 15 minutes, the procedure is repeated one more time.

DETAILED DESCRIPTION:
Endothelial dysfunction denotes abnormal contractile function of the inner lining of blood vessels. Endothelial dysfunction is associated with hypertension, hypercholesterolemia, atherosclerosis and diabetes and is an independent risk factor for cardiovascular disease. In normal physiology, endothelial cells synthesize and release factors that modulate blood vessel growth, inflammation, homeostasis, and vascular tone. Recently, endothelial dysfunction has been recognized as an early event in ischemia-reperfusion (IR) injury. IR injury causes damage to tissue and is important in many settings including acute coronary artery occlusions and cerebral ischemia. A model to examine the physiology of IR induced endothelial dysfunction and to test pharmacologic agents to prevent IR induced endothelial dysfunction is of paramount importance given the rise in cardiovascular and cerebrovascular disease. Recently in Protocol 06-H-0024, our group found that 20 minutes of ischemic stress causes no absolute endothelial dysfunction to the forearm using venous plethysmography to measure blood flow, despite numerous publications that support this model. We believe that the previously published data are based on a computational error resulting in an erroneous data interpretation (discussed in the introductory section of this proposal). Using NMR spectroscopy in protocol 06-H-0024 we have found that by adding exercise to exhaustion (usually 1 to 2 minutes of concentric exercise) to a 15-minute period of forearm ischemia results in a significantly more robust metabolic stress to the forearm, than 20 minutes of ischemia alone. Given the potential utilization of the restoration of endothelial function as a therapeutic strategy, we propose this pilot study to examine whether 15 minutes of ischemia with exercise to exhaustion (usually 1-2 minutes of concentric exercise) will cause transient IR dependent blunting of endothelial vasodilation as measured by venous plethysmography. In this study, an extension of Protocol 06-H-0024, we hypothesize that in human subjects the addition of concentric exercise to exhaustion, as a means to deplete high energy phosphate stores, will contribute to the development of transient endothelial dysfunction when performed in parallel with a 15-minute forearm ischemic stress. The establishment of a human system to enable the study of transient forearm vessel endothelial dysfunction will enable us to explore therapeutic interventions to protect against endothelial dysfunction.

ELIGIBILITY:
* ELIGIBILITY:

Up to 20 healthy volunteers will be screened in order to obtain 10 completed studies. All volunteer subjects will undergo screening with complete history, cardiovascular physical examination, electrocardiogram, blood collection for clinical chemistry routine analyses and complete blood count, cholesterol, fasting blood glucose, PT and PTT.

INCLUSION CRITERIA:

Subjects must be 18-45 years of age.

Subjects must be male.

Subject must be in good health.

Subject must complete a screening history and physical exam.

Subjects must provide informed, written consent for participation in this study.

EXCLUSION CRITERIA:

Subjects with a history of cardiac, pulmonary, peripheral vascular disease, coagulopathy, or any other disease predisposing to vasculitis or Raynaud's phenomenon.

Subjects with diabetes or mitochondrial disease.

Subjects with a history or evidence of present or past hypertension (blood pressure greater than 140/90 mmHg), hypercholesterolemia (LDL cholesterol greater than 160 mg/dL).

Subjects with abnormal EKG other than sinus bradycardia.

Subjects who have a history of smoking within three months.

Subjects with anemia (defined as hemoglobin less than 9 g/dL).

BMI greater than 30

No volunteer subject will be allowed to take any prescription medication. Vitamin supplements, herbal preparations, nutraceuticals or other alternative therapies must be stopped for two weeks prior to study and aspirin, tylenol and NSAIDs must also be discontinued two weeks prior to study.

Subjects with a blood pressure of less than 90/60 mmHg or mean arterial pressure (MAP) less than 70 mmHg on the study day will be excluded from the protocol.

Positive for HIV or Hepatitis B, C.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2007-03-26; Primary Completion 2009-02-11 (Actual); Study Completion 2009-02-11 (Actual)

PRIMARY OUTCOMES:
Change in vascular endothelial function.

SECONDARY OUTCOMES:
Assessment of systemic effects of this model system by assess contralateral arm blood flow and by assessing metabolic response to the combined exercise/ischemic stress.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rongen GA, Oyen WJ, Ramakers BP, Riksen NP, Boerman OC, Steinmetz N, Smits P. Annexin A5 scintigraphy of forearm as a novel in vivo model of skeletal muscle preconditioning in humans. Circulation. 2005 Jan 18;111(2):173-8. doi: 10.1161/01.CIR.0000151612.02223.F2. Epub 2004 Dec 27. PMID 15623546
- [Background] Kharbanda RK, Peters M, Walton B, Kattenhorn M, Mullen M, Klein N, Vallance P, Deanfield J, MacAllister R. Ischemic preconditioning prevents endothelial injury and systemic neutrophil activation during ischemia-reperfusion in humans in vivo. Circulation. 2001 Mar 27;103(12):1624-30. doi: 10.1161/01.cir.103.12.1624. PMID 11273988
- [Background] Broadhead MW, Kharbanda RK, Peters MJ, MacAllister RJ. KATP channel activation induces ischemic preconditioning of the endothelium in humans in vivo. Circulation. 2004 Oct 12;110(15):2077-82. doi: 10.1161/01.CIR.0000144304.91010.F0. Epub 2004 Oct 4. PMID 15466634